CLINICAL TRIAL: NCT02718105
Title: Maternal Killer Cell Immunoglobulin-like Receptors (KIR) and Fetal (Human Leukocyte Antigen) HLA-C Compatibility in ART-oocyte Donor Influences Live Birth Rate a Prospective Controlled Cohort Study
Brief Title: Maternal and Fetal Compatibility in Assisted Reproductive Technology (ART)-Oocyte Donor Influences Live Birth Rate
Status: Completed | Type: Observational
Sponsor: IVI Madrid (Other)
Responsible Party: Principal Investigator, Juan A Garcia-Velasco, PhD, IVI Madrid
Other Study IDs: 1512-MAD-067-JG
Record Dates: First submitted 2016-03-11; First posted 2016-03-24 (Estimated); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Infertility
Keywords: KIR HLA-C; ART
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genomic DNA will be obtained and will be studied in Professor Moffet laboratory in Cambridge (department of Pathologí, University of Cambridge) KIR typing including copi number and HLA-C loci will be performed as previously described (Hiby 2010, Jiang 2012). KIR haplotype regions will be defined by the presence of the following KIR genes: Cen-A/2DL3; Tel-A/3DL1 and 2DS4; Cen-B/2DL2 and 2DS2; Tel-B/2DS1 and 3DS1. The HLA-C ligands for KIRs will be divided into 2 groups: HLA-C1 and HLA-C2.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Receiver patients in donor oocyte -ART: Maternal and fetal compatibility KIR HLA-C determinations in ART -oocyte donor
  Interventions: Genetic: KIR HLAC determinations

INTERVENTIONS:
Genetic: KIR HLAC determinations — We will take blood samples for KIR HLA-C determinations.

SUMMARY:
Has the maternal KIR haplotype an impact in pregnancy, miscarriage and live birth rates per embryo transfer in donor oocytes -ART by paternal and oocyte donor HLA-C?

DETAILED DESCRIPTION:
The combination of maternal KIR haplotype and parental, donors HLA-C, could predict which couple can benefit for the selection of single embryo transfer (SET)/double embryo transfer (DET), or donor selection by HLA-C in ART, in order to increase the live birth rate (LBR)/cycle since HLA-C1/C1 donors are predicted to be safer and C2/C2 males or oocyte donors may be mor "dangerous" as identified by epidemiological studies

ELIGIBILITY:
Inclusion Criteria:

* BMI between 19 - 27 kg/m2
* Blastocyst embryo transfer previous.
* Normal karyotype, thrombophylic and immunological results.
* Normal clinical history, viral serology, hormonal analysis (TSH, T4, prolactin, estrogen, progesterone), spermiogram, sperm FISH and pelvic ultrasound results.

Exclusion Criteria:

* Pregnancy women.
* Psychiatric disorders.
* Uterus alterations.
* Polycystic ovary syndrome
* Genetic and autoimmune diseases.
* Infectious diseases.
* Corticoid and immunosuppressant treatments previous.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients undergoing an assisted reproductive treatment
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Compatibility maternal fetal KIR HLA-C | 2 years
  KIR haplotype regions will be defined by the presence of the following KIR genes: Cen-A/2DL3: Tel-A/3DL1 and 2DS4; Cen-B/2DL2 and 2DS2; Tel-B/2DS1 and 3DS1. The HLA-C ligands for KIRs will be divided into 2 groups: HLA-C1 and HLA_C2

CONTACTS AND LOCATIONS:
Overall Officials: Juan Antonio Garcia Velasco, PhD, Principal Investigator — IVI Madrid
Locations (1):
- Instituto Valenciano de Infertilidad, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No